CLINICAL TRIAL: NCT02433535
Title: Randomized Trial of Simvastatin for the Treatment of Severe Asthma
Brief Title: Trial of Simvastatin for the Treatment of Severe Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 522110; 522110-3 (Other: UC Davis)
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Severe Asthma
Keywords: severe asthma; simvastatin; allergic airway inflammation
MeSH Terms: conditions — Asthma | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Experimental): Simvastatin 40 mg daily will be given for 12 weeks.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): A placebo capsule will be given daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin is used to lower cholesterol, however, it also possess anti-inflammatory and immunomodulatory properties that may also alleviate allergic airway inflammation in asthma.
  Other Names: Zocor
  Arms: Simvastatin
Other: Placebo — A placebo pill will be given to the placebo group. There will be no detectible differences between study drug pill and placebo pill.
  Arms: Placebo

SUMMARY:
This purpose of this clinical trial is to determine if a statin drug, Simvastatin, added to inhaled corticosteroids and bronchodilators can reduce systemic and airway inflammation, improve lung function and symptoms, and reduce acute exacerbations in patients with severe asthma who are already on controller inhaler therapy.

This proposed investigator-initiated, single-center, early Phase II, cross-over, randomized clinical trial, titled "Randomized Trial of Simvastatin for the Treatment of Severe Asthma", will be conducted at the University of California, Davis Medical Center (UCDMC) in Sacramento, CA. This trial will evaluate Simvastatin for treatment of asthma in subjects with severe asthma (as defined by the American Thoracic Society (ATS)), who are already taking inhaler controller therapy. The investigators plan to enroll 24 patients with severe allergic asthma.

The investigators hypothesize that treatment with Simvastatin 40 mg (administered once daily) will not only improve indicators of airway and systemic allergic/Th2 inflammation, but will also reduce acute exacerbations and improve lung function. All patients will be on standard controller therapy including appropriate doses of inhaled corticosteroids and long-acting bronchodilators.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

1. statin-naïve adults >18 years old with the ATS definition of severe asthma,
2. on ICS and LABA,
3. confirmation of allergic asthma (serum IgE >100 kU/L, positive radioallergosorbent test (RAST) panel, and/or peripheral blood absolute eosinophil count of ≥700/mm3),
4. clinically stable for 4 weeks.

Exclusion Criteria:

1. baseline FEV1 <30% predicted,
2. current smokers or ex-smokers with >5 pack-years of smoking history,
3. pregnant women, nursing/lactating mothers, or women of childbearing potential who are actively attempting to become pregnant,
4. nasal or sinus surgery or trauma within 3 months of study participation,
5. ischemic heart disease,
6. liver disease, and
7. the concurrent use of the following medications (amiodarone, verapamil, diltiazem, gemfibrozil, cyclosporine, antifungal azoles (itraconazole, ketoconazole, or voriconazole), and danazol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Th2 gene expression in nasal epithelial cells. | Before and after 12 weeks of drug or placebo intervention.
  IL13, eotaxin-1,-2,-3, STAT6) by RT-PCR.
Exhaled nitric oxide (ENO) | Before and after 12 weeks of drug or placebo intervention.
  ENO will be measured using our NIOX-Mino portable NO analyzer.

SECONDARY OUTCOMES:
Acute Exacerbations | Before and after 12 weeks of drug or placebo intervention.
  Assessed as a rate per month.
Lung function | Before and after 12 weeks of drug or placebo intervention.
  FEV1, FVC, and FEV/FVC ratio.
Asthma symptom control score | Before and after 12 weeks of drug or placebo intervention.
  Asthma Control Test score (5 question survey).

CONTACTS AND LOCATIONS:
Locations (1):
- CTSC Clinical Research Center, Sacramento, California, United States